CLINICAL TRIAL: NCT03255330
Title: The Effect of Gabapentin Used as a Preemptive to the Emergence and Development Chronic Neuropathic Pain in Patients After Spinal Cord Trauma
Acronym: GabaNeuBol
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no participant enrolled
Sponsor: Masaryk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GNB-2015
Record Dates: First submitted 2017-08-15; First posted 2017-08-21 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Chronic Pain Due to Trauma; Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Gabapentin; Dipyrone; Tramadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm G1800 (Experimental): administration of gabapentin with a gradual increasing dose of up to 1800 mg / day
  Interventions: Drug: Gabapentin
- G0 (Active Comparator): Standardized medical treatment of central neuropathic pain: metamizole, tramadol
  Interventions: Drug: Metamizol; Drug: Tramadol

INTERVENTIONS:
Drug: Gabapentin — Gabapentin will be given approximately 3 months until no chronic neuropathic pain is present
  Other Names: Gabapentinum
  Arms: Arm G1800
Drug: Metamizol — Standardized treatment
  Arms: G0
Drug: Tramadol — Standardized treatment
  Arms: G0

SUMMARY:
Study of the effect of gabapentin used as a preemptive to the emergence and development chronic neuropathic pain in patients after spinal cord trauma

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age 18 - 65 years
2. Signed written informed consent
3. Patients after complete/non-complete spinal lesion, after surgery
4. Patients with spinal cord trauma caused mechanically demanding (due a injury of a bone fragment, a disk, a translation spinal canal)
5. Patient willing and able to comply with the study protocol
6. Male and females with a highly effective method of birth control plus an additional barrier method

Exclusion Criteria:

1. Patients with spinal cord lesion ischemic etiology
2. Pregnant women, nursing or childbearing age with a positive pregnancy test input
3. Patients unable or unwilling to comply with the study protocol
4. Acute pancreatitis in 1 year from the start of the study
5. Chronic pancreatitis in the case history
6. Active or uncontrolled infectious diseases
7. Hypersensitivity to any component of the investigational product
8. Active autoimmune disease
9. Serious neurological disease with the incidence chronic neuropathic pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Assessment the analgesic effect of gabapentin | in 3 months after initiation of the gabapentin treatment
  The decrease of the incidence of chronic neuropathic pain in 3 months after initiation of the gabapentin treatment in 3 months after initiation of the gabapentin treatment

SECONDARY OUTCOMES:
The decrease of the incidence of chronic neuropathic pain | in 6., 9. and 12. months after initiation of the gabapentin treatment
  The decrease of the incidence of chronic neuropathic pain in 6., 9. and 12. months after initiation of the gabapentin treatment
The number of painful episodes | in 3., 6., 9. and 12. months after initiation of the gabapentin treatment
  The number of painful episodes requiring treatment of rescue medication (in 3., 6., 9. and 12. months after initiation of the gabapentin treatment)
The decrease of the consumption of rescue medication | in 3., 6., 9. and 12. months after initiation of the gabapentin treatment
  The decrease of the consumption of rescue medication in 3., 6., 9. and 12. months after initiation of the gabapentin treatment
Absolute and percentage change in average pain | in 3., 6., 9. and 12. months
  Absolute and percentage change in average pain after initiation of therapy with gabapentin (baseline) in 3., 6., 9. and 12. months
Quality of life | in week 1, 3., 6., 9. and 12. months after initiation of the gabapentin treatment
  Quality of life, assessment of neurological pain and psychological state measured by questionnaires PainDETECT, SQUALA and SCL-R

CONTACTS AND LOCATIONS:
Locations (1):
- Fakultní nemocnice Brno, Brno, Czechia